CLINICAL TRIAL: NCT06288048
Title: EFECTIVIDAD DE LA TERAPIA EN ESPEJO EN EL DOLOR POSTPUNCIÓN DE PUNTOS GATILLO MIOFASCIALES [EFFECTIVENESS OF MIRROR THERAPY ON POST-PUNCTURE PAIN OF MYOFASCIAL TRIGGER POINTS]
Brief Title: Effect of Mirror Therapy on Post-Needling Pain Following Deep Dry Needling of Myofascial Trigger Point in Lateral Elbow Pain
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidad Europea de Canarias (Other)
Responsible Party: Principal Investigator, Sebastian Eustaquio Martin Perez, Full-Time Professor, Universidad Europea de Canarias
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23/107-EC X TFM 07/03/2023
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Lateral Elbow Pain
Keywords: Mirror Therapy; Dry Needling; Post-Needling Pain; Myofascial Trigger Point
MeSH Terms: interventions — dendrin; Acupressure; D-4-chloro-17 beta-hydroxy-3-oxo-17 alpha-methylandrosta-1,4-diene

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Allocation and data assessor were blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep Dry Needling (DDN), Ischemic Compression, Cold Spray with Stretching + MFT (Experimental): The intervention protocol in this study will target individuals experiencing Post-needling pain associated with lateral elbow pain. It will comprise a series of treatments including Deep Dry Needling (DDN) focused on the proximal third of the m. Brachioradialis (BR), was conducted with the patient seated and the therapist positioned on the same side as the needle insertion. Following DDN, ischemic compression (IC) will be applied using a sphygmomanometer on the seated subject's arm, along with three applications of cold spray synchronized with m. Brachioradialis (BR) stretching. The intervention will conclude with Mirror Therapy (MFT), where the patient will face a mirror covering the punctured side at a 45-degree angle for proper hand visualization, engaging in hand exercises and wrist movements while observing their reflection.
  Interventions: Procedure: Experimental: Deep Dry Needling (DDN), Ischemic Compression, Cold Spray with Stretching + MFT
- Deep Dry Needling (DDN), Ischemic Compression, Cold Spray with Stretching (Active Comparator): The intervention protocol in this study will target individuals experiencing Post-needling pain associated with lateral elbow pain. It will comprise a series of treatments including Deep Dry Needling (DDN) focused on the proximal third of the m. Brachioradialis (BR), conducted with the patient seated and the therapist positioned on the same side as the needle insertion. Following DDN, ischemic compression (IC) will be applied using a sphygmomanometer on the seated subject's arm, along with three applications of cold spray synchronized with m. Brachioradialis (BR) stretching. The intervention will not conclude with Mirror Therapy (MFT).
  Interventions: Procedure: Deep Dry Needling (DDN), Ischemic Compression, Cold Spray with Stretching

INTERVENTIONS:
Procedure: Experimental: Deep Dry Needling (DDN), Ischemic Compression, Cold Spray with Stretching + MFT — Experimental:
  Target: Proximal third of m. Brachioradialis (BR) Patient position: Seated Therapist position: Same side as needle insertion Needle insertion direction: Lateral-to-medial towards clinician's finger Needle type: AguPunt® Barcelona, Spain Technique: Seek three local twitch responses in m. Brachioradialis (BR) Alternative for no responses: 10 needle insertions and withdrawals at 1 Hz frequency
  Ischemic Compression (IC):
  Applied using sphygmomanometer on seated subject's arm Pressure: Increased until ischemic pain (approx. 200 mmHg) Duration: Maintained for 90 seconds
  Combined with three applications of Cryos Phyto Performance 400 ml cold spray synchronized with m. Brachioradialis (BR) stretching:
  Stretching: Passive sustained mobilization with elbow extension and forearm pronation for 10 seconds
  Mirror Therapy (MFT):
  Setup: Patient seated with forearms resting on bed Mirror: 35 x 35 cm, covering punctured side at 45-degree angle for hand visualization
  Arms: Deep Dry Needling (DDN), Ischemic Compression, Cold Spray with Stretching + MFT
Procedure: Deep Dry Needling (DDN), Ischemic Compression, Cold Spray with Stretching — The intervention protocol in this study will target individuals experiencing Post-needling pain associated with lateral elbow pain. It will comprise a series of treatments including Deep Dry Needling (DDN) focused on the proximal third of the m. Brachioradialis (BR), conducted with the patient seated and the therapist positioned on the same side as the needle insertion. Following DDN, ischemic compression (IC) will be applied using a sphygmomanometer on the seated subject's arm, along with three applications of cold spray synchronized with m. Brachioradialis (BR) stretching. The intervention will not conclude with Mirror Therapy (MFT).
  Arms: Deep Dry Needling (DDN), Ischemic Compression, Cold Spray with Stretching

SUMMARY:
The goal of this randomized, controlled pilot trial is to investigate the immediate effects of incorporating Mirror Visual Feedback Therapy (MFT) on pain sensitivity and motor performance in individuals experiencing Post-needling pain associated with lateral elbow pain. The main questions it aims to answer are:

* Does incorporating Mirror Visual Feedback Therapy reduce Post-needling pain intensity?
* Does incorporating Mirror Visual Feedback Therapy improve pressure pain threshold?
* Does incorporating Mirror Visual Feedback Therapy improve maximum grip strenght?

Participants will be asked to undergo pre- and post-treatment evaluations, which include assessments of Post-needling pain intensity, pressure pain threshold, two-point discrimination threshold, and maximum hand grip strength.

Participants in the Experimental Group will receive Deep Dry Needling in the m. Brachioradialis, Ischemic Compression, Cold Spray, Stretching, and Mirror Visual Feedback Therapy. Those in the Control Group will not receive Mirror Visual Feedback Therapy.

Researchers will compare the Experimental Group to the Control Group to see if the incorporation of Mirror Visual Feedback Therapy results in a reduction in Post-needling pain intensity and improvement in pressure pain threshold.

DETAILED DESCRIPTION:
This randomized, controlled pilot trial aims to investigate the immediate effects of incorporating Mirror Visual Feedback Therapy (MFT) on pain sensitivity and motor performance in individuals experiencing Post-needling pain associated with lateral elbow pain. The study will enroll a total of 49 participants, with 23 females and 26 males, who will be randomly allocated to either the Experimental Group or the Control Group. The Experimental Group will receive Deep Dry Needling in the m. Brachioradialis, Ischemic Compression, Cold Spray, Stretching, and Mirror Visual Feedback Therapy, while the Control Group will not receive Mirror Visual Feedback Therapy. This random allocation is intended to minimize bias and enhance the internal validity of the study.

Pre- and post-treatment evaluations will include assessments of Post-needling pain intensity, pressure pain threshold, two-point discrimination threshold, and maximum hand grip strength. Intergroup analysis will be conducted to determine if there is a statistically significant reduction in Post-needling pain intensity favoring the Experimental Group. Additionally, intragroup analysis will assess whether there are significant improvements in pressure pain threshold solely within the Experimental Group following the intervention.

The findings of this study may suggest a potential benefit of integrating MFT into treatment protocols for individuals with lateral elbow pain experiencing Post-needling discomfort. However, further research will be necessary to fully elucidate the clinical implications of these findings and their applicability in healthcare settings.

ELIGIBILITY:
Inclusion Criteria:

* Individuals males and females aged 18 years or older
* Individuals suffering from lateral elbow myofascial pain diagnosed by either a GP or physical therapist
* for less than 3 months
* lacking a history of severe trauma
* Individuals not having any prior exposure to Dry Needling treatment
* Individuals not currently using relevant medications

Exclusion Criteria:

* Individuals under the age of 18
* Individuals not diagnosed with lateral elbow myofascial pain by either a GP or physical therapist
* Individuals experiencing lateral elbow myofascial pain for more than 3 months
* Individuals with a history of severe trauma to the affected area
* Individuals who have previously undergone Dry Needling treatment for their lateral elbow myofascial pain
* Individuals currently using medications relevant to the treatment of lateral elbow myofascial pain

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-03-07 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | From before and after the intervention until the conclusion of treatment at the 1-hour.
  Pain intensity refers to the subjective level of discomfort or suffering experienced by an individual due to pain. It will be measured in Visual Analogue Scale (VAS).
Pain pressure threshold | From before and after the intervention until the conclusion of treatment at the 1-hour.
  The pain pressure threshold refers to the amount of pressure or force applied to a specific area of the body before the sensation of pain is experienced. It is commonly used in medical evaluations to assess pain sensitivity and tolerance. It will be measured in PPT (Kg/cm2)
Two-point discrimination threshold | From before and after the intervention until the conclusion of treatment at the 1-hour.
  The two-point discrimination threshold refers to the ability of an individual to perceive two separate points of contact on the skin as distinct from a single point. It will be measured in 2-point discriminator 12-1480 skin caliper Baseline®.
Maximum hand grip strength | From before and after the intervention until the conclusion of treatment at the 1-hour.
  Maximum hand grip strength refers to the maximum force that an individual can exert when squeezing an object with their hand muscles. It will be measured JAMAR® Hand Dynamometer J00105.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea de Canarias, La Orotava, Santa Cruz De Tenerife, Spain

IPD SHARING:
Plan to Share IPD: No
Results should not be shared, although they will be available to reviewers upon request.

REFERENCES:
- [Result] Martin-Pintado-Zugasti A, Mayoral Del Moral O, Gerwin RD, Fernandez-Carnero J. Post-needling soreness after myofascial trigger point dry needling: Current status and future research. J Bodyw Mov Ther. 2018 Oct;22(4):941-946. doi: 10.1016/j.jbmt.2018.01.003. Epub 2018 Jan 17. PMID 30368339